CLINICAL TRIAL: NCT05234957
Title: Symmetric Versus Asymmetric Bilateral Lateral Rectus Recession in Management of Basic Intermittent Exotropia With Ocular Dominance
Brief Title: Symmetric vs Asymmetric BLR Recession in Management of Basic IXT With Ocular Dominance
Acronym: IXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Mohamed Fathy Farid, Professor, Benha University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RC1-1-2022
Record Dates: First submitted 2022-01-20; First posted 2022-02-10 (Actual); Results first posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-10

CONDITIONS: Intermittent Exotropia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Active Comparator): Symmetric bilateral lateral rectus recession (S-BLR). The amount of bilateral lateral rectus recession is equally divided between both eyes.
  Interventions: Procedure: Bilateral Lateral Rectus Recession
- Group 2 (Active Comparator): Asymmetric bilateral lateral rectus recession (A-BLR). The amount of bilateral lateral rectus recession is asymmetrically divided between both eyes, with 2mm more recession in the non-dominant eye.
  Interventions: Procedure: Bilateral Lateral Rectus Recession

INTERVENTIONS:
Procedure: Bilateral Lateral Rectus Recession — Symmetric bilateral lateral rectus muscle recession involves equal recession of both lateral rectus muscles. Asymmetric bilateral lateral rectus muscle recession involves recession of the lateral rectus muscle by 2mm more in the non-dominant eye.

SUMMARY:
The study aims to investigate ocular motor and sensory outcomes of two different strategies of lateral rectus recession; symmetric and asymmetric, in management of basic type intermittent exotropia with ocular dominance.

DETAILED DESCRIPTION:
Surgical management of basic -type intermittent exotropia with a dominant eye is controversial. Some surgeons do traditional symmetrical bilateral lateral rectus recession, while other perform unilateral recess-resect procedure in the non-dominant eye. The aim of this study is to investigate the effect of two different strategies of bilateral lateral rectus recession; symmetrical recession in which the amount of recession is equally divided between both eyes, and asymmetrical recession, in which the amount of recession is 2mm more in the non-dominant. Outcome measures include ocular deviation at distant and near fixation, sensory status and complications.

ELIGIBILITY:
Inclusion Criteria:

* Basic-type intermittent exotropia
* Simulated distant-type intermittent exotropia

Exclusion Criteria:

* Alternating basic-type intermittent exotropia (no ocular dominance)
* Distant-type intermittent exotropia
* Convergence-insufficiency type intermittent exotropia
* Constant exotropia
* Sensory exotropia
* Deep amblyopia
* Paralytic or restrictive exotropia
* Previous extraocular muscle surgery

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-04-17 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Farid, MD, Principal Investigator — Benha University
Locations (1):
- Benha University, Banhā, Qalyubiyya, Egypt

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.85 (5.42) | 8.75 (5.48) | 9.3 (5.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 20 | 20 | 40
Best Corrected Visual Acuity Right Eye (BCVA/OD) [Mean (Standard Deviation); unit: logMAR] | 0.05 (0.06) | 0.02 (0.06) | 0.03 (0.06)
Best Corrected Visual Acuity Left Eye (BCVA/OS) [Mean (Standard Deviation); unit: logMAR] | 0.06 (0.09) | 0.03 (0.07) | 0.05 (0.08)
Spherical Equivalent Refractive Error Right Eye (SE/0D) [Mean (Standard Deviation); unit: diopter] | -0.03 (0.74) | -0.41 (1.3) | -0.22 (1.08)
Spherical Equivalent Refractive Error Left Eye (SE/OS) [Mean (Standard Deviation); unit: diopter] | 0.1 (0.89) | -0.55 (2.18) | -0.22 (1.68)
Ocular Dominance Right Eye [Count of Participants; unit: Participants] | 16 | 12 | 28
Ocular Dominance Left Eye [Count of Participants; unit: Participants] | 4 | 8 | 12
preoperative distant deviation [Mean (Standard Deviation); unit: prism diopter] | 36.25 (9.01) | 32.25 (6.97) | 34.25 (8.2)
preoperative near deviation [Mean (Standard Deviation); unit: prism diopter] | 36.25 (10.1) | 32.75 (7.51) | 34.5 (8.97)
Fusion [Count of Participants; unit: Participants] — Assessment of binocular fusion by using Worth's dot test. Patients who can fuse are termed (positive fusion), and patients who can not fuse are termed (absent fusion).
  Participants
    positive fusion | 5 | 6 | 11
    absent fusion | 15 | 14 | 29
preoperative stereopsis [Mean (Standard Deviation); unit: second of arc] | 251 (171.4) | 263 (172.4) | 257 (169.8)

OUTCOME MEASURES:

1. Primary Outcome: Ocular Alignment at Distant Fixation
Description: ocular alignment in prism diopter (PD) at distant fixation (6 meter) is measured using alternate prism and cover test (APCT) while patient wears refractive correction.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: prism diopter
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 20 | 20
prism diopter | 5.8 (5.54) | 1.1 (4.7)

2. Primary Outcome: Ocular Alignment at Near Fixation
Description: ocular alignment in prism diopter (PD) at near fixation (1/3 meter) is measured using alternate prism and cover test (APCT) while patient wears refractive correction.
Time Frame: one year
Measure: Mean (Standard Deviation); unit: prism diopter
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 20 | 20
prism diopter | 6.6 (5.52) | 3.5 (6.19)

3. Secondary Outcome: Sensory Status (Stereopsis)
Description: ocular sensory status (stereopsis) is assessed using Titmus fly test and is recorded as seconds of arc.
Time Frame: one year
Population: Stereopsis
Measure: Mean (Standard Deviation); unit: second of arc
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 20 | 20
second of arc | 124 (81.3) | 119.5 (54.2)

4. Secondary Outcome: Sensory Status (Fusion)
Description: Fusion is assessed using Worth 4-dot test, and is documented as present (positive fusion) or absent (absent fusion).
Time Frame: one year
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 20 | 20
Participants
  positive fusion | 5 | 6
  absent fusion | 15 | 14

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 8/20 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (N=20) | Group 2 (N=20)
undercorrection/recurrence (Eye disorders) | 8 | 4 — postoperative deviation equal or greater than 10 prism diopter exotropia/phoria at distant and/or near fixation.
overcorrection (Eye disorders) | 0 | 1 — postoperative deviation equal or greater than 10 prism diopter esotropia/phoria at distant and/or near fixation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT05234957/Prot_SAP_000.pdf